CLINICAL TRIAL: NCT01404143
Title: Comparison of Two Methods of Subscapularis Management in Shoulder Arthroplasty: Tenotomy Versus Peel: A Multicenter, Randomized Controlled
Brief Title: Comparison of Two Methods of Subscapularis Management in Shoulder Arthroplasty: Tenotomy Versus Peel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: St. Joseph's Health Care London (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-352
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Subscapularis Injury

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subscapularis Tenotomy (Active Comparator): This treatment group will undergo a technique that involves division of the tendon to gain access to the shoulder.
  After the deltopectoral approach is completed, the subscapularis tendon will be tenotomized one centimeter medial to its insertion on the lesser tuberosity.
  Interventions: Procedure: Subscapularis Tenotomy
- Subscapularis Peel (Experimental): This treatment group will use a technique that involves elevation of the tendon off the bone in order to gain access to the shoulder.The subscapularis will be elevated from the lesser tuberosity.
  Interventions: Procedure: subscapularis peel

INTERVENTIONS:
Procedure: Subscapularis Tenotomy — After the deltopectoral approach is completed, the subscapularis tendon will be tenotomized one centimeter medial to its insertion on the lesser tuberosity. The tendon will be tagged for later repair. Repair will take place with a combination of transosseous sutures (3) placed in a mattress configuration through the area of exposed lesser tuberosity. In addition, a soft tissue tendon to tendon repair will be carried out using figure-8 stitches using #2 (heavy) non-absorbable suture (Ticron).
  Arms: Subscapularis Tenotomy
Procedure: subscapularis peel — The subscapularis will be elevated from the lesser tuberosity. The tendon will be tagged with stay sutures for later reattachment (3 sutures in mattress configuration). Reapproximation will take place with three non-absorbable mattress sutures placed in a trans-osseous fashion through the bicipital groove, exiting the greater tuberosity and tied over a 4-hole mini-fragment plate.
  Arms: Subscapularis Peel

SUMMARY:
What is the difference in subscapularis strength between two different methods of subscapularis mobilization: incision of the tendon (tenotomy) versus peel.

It is the investigators' hypothesis that a peel of the subscapularis will result in greater strength, a higher healing rate, and a greater improvement in shoulder function and quality of life following shoulder replacement.

DETAILED DESCRIPTION:
The primary research question is to determine the difference in subscapularis strength between two different methods of subscapularis mobilization in shoulder arthroplasty: intra-substance division of the tendon "tenotomy" versus direct detachment of the subscapularis tendon from its insertion on the lesser tuberosity "the peel". The primary outcome is strength as measured by a hand-held dynamometer in the belly-press position at one-year post operative. Secondary research questions include determination of the difference in disease specific quality of life between patients who undergo a subscapularis tenotomy versus subscapularis peel, as measured by the Western Ontario Osteoarthritis of the Shoulder Index (WOOS), Constant score and the ASES score at one year post-operatively. Finally, the healing rate of the subscapularis, as measured by ultrasound at 1 year post-operative will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Imaging, and intra-operative findings confirming advanced humeral head cartilage loss, and/glenoid cartilage loss.
* Ability to understand and adhere to rehab protocols and testing procedure
* Persistent pain and functional disability for at least 6 months and failure of 6 months of conservative treatment
* surgical arthroplasty patients

Exclusion Criteria:

* Active joint of systemic infection
* Significant muscle paralysis
* Rotator cuff tear arthropathy
* Pregnancy
* Charcot's arthropathy
* Major medical illness ( life expectancy less then 1 year or unacceptably high operative risk)
* Patients unable to provide informed consent due to language barrier or mental status
* Unable to speak or read English/French
* Psychiatric illness that precludes informed consent
* Patients unwilling to be followed for the duration of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
What is the difference in subscapularis strength between two different methods of subscapularis mobilization: incision of the tendon (tenotomy) versus peel | 12 months
  What is the difference in subscapularis strength between two different methods of subscapularis mobilization: incision of the tendon (tenotomy) versus peel, as measured by a hand-held dynamometer in the belly-press position at one year post operative?

SECONDARY OUTCOMES:
Quality of life as measured by WORC, ASES and Constant | 12 months
  1. What is the difference in disease specific quality of life between patients who undergo a subscapularis tenotomy versus peel, as measured by the Western Ontario Osteoarthritis of the Shoulder Index (WOOS) at one year post-operatively in patients who undergo shoulder arthroplasty?
  2. What is the difference in outcome as measured by the Constant score and the ASES score, at one year post operatively?
  3. What are the healing rates, as measured by ultrasound at 1 year post-operative?

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lapner, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided